CLINICAL TRIAL: NCT00822471
Title: Feasibility and Impact of of "ABC's of Diabetes" Self Management Education (DSME) Program for African Americans at an Urban Public Library on A1C, Lipid Lowering Agent Prescriptions and Emergency Department Visits
Brief Title: Feasibility and Impact of "ABCs of Diabetes" Self-Management Education Program at an Urban Public Library
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Medstar Diabetes Institute; (Unknown); American Diabetes Association (Other); Bayer (Industry); CareFirst BlueCross Blue Shield; (Unknown); District of Columbia, Department of Health Block Grants Program; (Unknown); Charles and Mary Latham Trust Fund; (Unknown); Eli Lilly and Company (Industry); Hewlett-Packard (Industry); Meltzer Entities; (Unknown); NBC Washington (Other); Novo Nordisk A/S (Industry); Aventis Pharmaceuticals (Industry); Takeda Pharmaceuticals North America, Inc. (Industry); Pfizer (Industry)
Responsible Party: Principal Investigator, Michelle Magee, Professor of Medicine, Georgetown University School of Medicine, Medstar Health Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2002-288
Record Dates: First submitted 2009-01-12; First posted 2009-01-14 (Estimated); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Diabetes; Cardiovascular Disease
Keywords: Diabetes; Self-Management Education; Library; Emergency Department Visits; African American; CVD prevention; Prevention; Uncontrolled diabetes
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diabetes Self-Management Education (Other): Education intervention with historic self-controls.
  Interventions: Behavioral: Diabetes Self-Management Education

INTERVENTIONS:
Behavioral: Diabetes Self-Management Education — DSME intervention consisting of two interactive 2-1/2 hour classes taught by a diabetes educator focusing on the "ABCs of diabetes" and training in how to talk to your doctor.

SUMMARY:
A concise diabetes self-management education (DSME) program on the "ABCs of Diabetes" will be placed in an urban public library to assess the feasibility of using this community setting for the delivery of health care education in an urban African American population. Impact on knowledge of, prescriptions for, and control of blood sugar (A1C), blood pressure (BP) and LDL cholesterol (LDL-C)before and after participation in the program will be assessed. We will also examine the frequency of emergency department (ED) visits and hospitalizations for uncontrolled diabetes at 6 months post-DSME intervention.

DETAILED DESCRIPTION:
A free, community-based Diabetes Learning Center was placed in a public library. Adults with diabetes (N=360) consented to participate in this prospective cohort study with historic self-controls. The small group, interactive DSME (two 2-1/2 hour classes) focused on improving CVD risk factors and enabling communication with the primary care physician. Knowledge, prescriptions, diabetes-related testing and clinical outcomes were assessed.

"ABCs of Diabetes" DSME Program

Class #1: A1C, Aspirin & Blood Pressure

A. Curriculum Content Areas:

* What is diabetes?
* A1C and blood glucose targets
* Diabetes medications
* Hypoglycemia
* Managing Blood Pressure
* Taking your medications
* Preventing vascular complications
* Monitoring your diabetes health
* "How to Talk to your Doctor"

B. Education strategies & tools

* Role playing from "How To Talk to Your Doctor"
* Ask for test results and how to get to targets
* Prompts to schedule appointments for ADA recommended exams, tests and discuss diabetes with primary care provider

Class #2 Cholesterol and Meal Planning

A. Curriculum Content Areas:

* Managing cholesterol
* Diet, exercise & weight management
* Cholesterol medications
* Smoking cessation
* Family Meal Planning:

consistent carbohydrate

* heart healthy meals

B. Education strategies & tools

* View "Cut the Fat Back" video†
* Interactive portion size & meal planning strategies
* Prompts to query PCP for LDL-C results;
* Flyers with questions to focus PCP on ADA goals † Produced by the Health Promotion Council, Philadelphia PA hpcpa@phmc.org

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Diabetes Mellitus, type 1 or type 2 for at least one month prior to taking the first educational class.
2. 18 years old or older.
3. Females and Males
4. All ethnic groups.
5. Must be able to read and speak English.
6. Must be willing to sign informed consent to participate in the research component of the program.
7. Plan on living in the District of Columbia for the next 6 to 8 months.
8. Willing to attend 2 core interactive education sessions within a 6-week period.
9. Willing to have a fingerstick performed to obtain blood for A1C and cholesterol determinations prior to and 6 months after completion of the educational sessions.
10. Willing to attend both a pre- and a post-study outcomes data collection visit, each of which will last approximately 1 - 1 ½ hours.
11. Ability and willingness to adhere to all study requirements.
12. Participant must have active health insurance coverage or self pay and have regular visits to their primary care physician. Interested parties who do not have health insurance will be referred to DHHS for assistance in applying for Medicare or Medicaid when applicable.
13. Have access to telephone in residence to receive reminder calls for up upcoming visits.

Exclusion Criteria:

1. Pregnancy.
2. Non-English speaking.
3. Untreated mental illness.
4. History of substance abuse or alcohol abuse in the past 12 months.
5. Individuals participating in a drug research study.
6. Presence of concomitant condition or circumstances which, in the opinion of the investigator, could interfere with participation in the study, glycemic control or interpretation of the data collected. (e.g. active malignance; HIV/AIDS)
7. Chronic concomitant use of oral steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2003-01; Primary Completion 2005-01 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Improvement in the percent of subjects correctly identifying guideline-recommended treatment targets for the "ABC's of Diabetes", where A = A1C < 7%; B = BP <130/80mmHg and; and C = LDL-C < 100mg/dl. | 6 months following program completion

SECONDARY OUTCOMES:
increase the percentage of subjects taking medications for A1C, BP and LDL-C management and aspirin; | 6 months following DSME program completion
increase scores on the diabetes self-efficacy scale (DES); | 6 months following DSME program completion
increase percentage of patients with A1C, BP and LDL-C at recommended targets; | 6 months following program completion
Decrease the percentage of participants with self-reported ED visits and hospitalizations for severe hypoglycemia and hyperglycemia. | 6 months following DSME program completion

CONTACTS AND LOCATIONS:
Overall Officials: Michelle F. Magee, MD, LRCPSI, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States